CLINICAL TRIAL: NCT04940676
Title: Oral Administration or Nasal Feeding of Huzhangxiefei Decoction for Treatment in Sepsis Induced Acute Lung Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-21-005
Record Dates: First submitted 2021-06-24; First posted 2021-06-25 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-06

CONDITIONS: Acute Lung Injury; Sepsis
Keywords: acute lung injury; sepsis; Chinese Traditional Medicine; Chinese Herbal Drugs; acute respiratory distress syndrome
MeSH Terms: conditions — Acute Lung Injury; Sepsis; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huzhangxiefei Decoction (Active Comparator): Huzhangxiefei Decoction, 50ml, Oral Administered or Nasal Feeding 5 minutes after breakfast and dinner for 7 days
  Interventions: Drug: Huzhangxiefei Decoction
- 10% Huzhangxiefei Decoction (Placebo Comparator): 10% Huzhangxiefei Decoction, 50ml, Oral Administered or Nasal Feeding of 5 minutes after breakfast and dinner for 7 days
  Interventions: Drug: 10% Huzhangxiefei Decoction

INTERVENTIONS:
Drug: Huzhangxiefei Decoction — Huzhangxiefei Decoction, 50ml, Oral Administered or Nasal Feeding 5 minutes after breakfast and dinner for 7 days
  Arms: Huzhangxiefei Decoction
Drug: 10% Huzhangxiefei Decoction — 10% Huzhangxiefei Decoction, 50ml, Oral Administered or Nasal Feeding 5 minutes after breakfast and dinner for 7 days
  Arms: 10% Huzhangxiefei Decoction

SUMMARY:
Hypothesis 1A: Oral Administration or Nasal Feeding of Huzhangxiefei Decoction will significantly attenuate sepsis-induced systemic organ failure as measured by overall response rate.

Hypothesis 1B: Oral Administration or Nasal Feeding of Huzhangxiefei Decoction will attenuate sepsis-induced lung injury as assessed by the respiratory rate and oxygenation index.

Hypothesis 1C: Oral Administration or Nasal Feeding of Huzhangxiefei Decoction will attenuate sepsis-induced lung injury as assessed by chest x-ray scale score, Chinese Medicine scale score.

Hypothesis 1D: Oral Administration or Nasal Feeding of Huzhangxiefei Decoction will attenuate biomarkers of inflammation (C-Reactive Protein, Procalcitonin), vascular injury (Thrombomodulin, Angiopoietin-2), alveolar epithelial injury (Receptor for Advanced Glycation Products), while inducing the onset of a fibrinolytic state (Tissue Factor Pathway Inhibitor).

DETAILED DESCRIPTION:
Huzhangxiefei Decoction is a prescription formulated by a professional doctor of traditional Chinese medicine

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suspected or proven infection, and be accompanied by at least 1 criterion for sepsis-induced organ dysfunction, and meet all 5 criteria for Acute Respiratory Distress Syndrome (ARDS).

Suspected or proven infection: (e.g., thorax, urinary tract, abdomen, skin, sinuses, central venous catheters, and central nervous system).

The presence of sepsis associated organ dysfunction: (any of the following thought to be due to infection): Sepsis associated hypotension (systolic blood pressure (SBP) < 90 mm Hg or an SBP decrease > 40 mm Hg unexplained by other causes or use of vasopressors for blood pressure support (epinephrine, norepinephrine, dopamine =/> 5mcg, phenylephrine, vasopressin); Arterial hypoxemia (PaO2/FiO2 < 300) or supplemental O2 > 6LPM; Lactate > upper limits of normal laboratory results; Urine output < 0.5 ml/kg/hour for > two hours despite adequate fluid resuscitation; Platelet count < 100,000 per mcL; Coagulopathy (INR > 1.5); Bilirubin > 2 mg/dL; Glasgow Coma Scale < 11 or a positive CAM ICU score.

ARDS characterized by all the following criteria Lung injury of acute onset, within 1 week of an apparent clinical insult and with progression of respiratory symptoms Bilateral opacities on chest imaging not explained by other pulmonary pathology (e.g. pleural effusions, lung collapse, or nodules) Respiratory failure not explained by heart failure or volume overload Decreased arterial PaO2/FiO2 ratio ≤ 300 mm Hg Minimum PEEP of 5 cmH2O (may be delivered noninvasively with CPAP to diagnose mild ARDS

Exclusion Criteria:

* inability to obtain consent;
* age < 18 years;
* pregnancy or breast feeding;
* moribund patient not expected to survive 24 hours;
* for patients with chronic liver insufficiency, renal insufficiency, blood system disease, etc., it is impossible to judge that the organ insufficiency occurred after this infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) Score | up to 7 days
  SOFA is a single score based on patient status of five different biological systems: respiratory, cardiovascular, coagulation, renal, and neurological. Scores range from 0 to 24 with higher scores indicated worse status
C-Reactive Protein at Study Hours 0, 96, 168 When Compared to Placebo | up to 168 hours
  C-Reactive Protein at Study Hours 0, 96, 168 When Compared to Placebo
Oxygenation Index (FiO2 x Mean Airway Pressure/PaO2) at Study Hour 0, 96, 168 if Still Intubated in Oral Administration or Nasal Feeding of Huzhangxiefei decoction Patient Compared to Placebo | up to 168 hours
  Oxygenation Index (FiO2 x Mean Airway Pressure/PaO2) at Study Hour 0, 96, 168 if Still Intubated in Oral Administration or Nasal Feeding of Huzhangxiefei decoction Patient Compared to Placebo
overall response rate | up to 7 days
  Overall response rate=(the number of marked response patients+the number of moderate response)/the number of all patients within group
  Four criteria were established as follows:
  1. RR(d1)-RR(d7)≥5 breaths per minute or 12 breaths per minute≤RR(d7)≤20breaths per minute
  2. OI(d7)-OI(d1)≥50mmHg
  3. [CXSS(d1)-CXSS(d7)]/CXSS(d1)≥10%
  4. CMSS(d1)-CMSS(d7)≥3 points Marked response: three or four criteria of the above are met Moderate response：two criteria of the above are met No response: none or only one criterion of the above is met
  RR refers to respiratory rate, breaths per minute OI refers to oxygenation index, mmHg CXSS refers to chest x-ray scale score CMSS refers to Chinese Medicine scale score

SECONDARY OUTCOMES:
Ventilator Free Days to Day 28 | Up to Day 28
  Ventilator Free Days to Day 28
ICU-free Days at Day 28 | Up to Day 28
  ICU-free Days at Day 28
All Cause Mortality to Day 28 | Up to Day 28
  All Cause Mortality to Day 28
Hospital-free Days at Day 60 | Up to Day 60
  Hospital-free Days at Day 60
Procalcitonin at Study Hour 0, 96, 168 | Up to hour 168
  Procalcitonin at Study Hour 0, 96, 168
Tissue Factor Pathway Inhibitor at Study Hour 0, 96, 168 | Up to hour 168
  Tissue Factor Pathway Inhibitor at Study Hour 0, 96, 168
Oxygenation Score: Pressure | Up to hour 168
  Oxygenation as measure by the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2). Scores range from 100 to 300 with lower values indicating more worse outcomes
Coagulation | Up to hour 168
  Coagulation as measured by Platelets per unit of blood. Scores range from less than 20 to more than 150. Lower scores indicate worse outcomes
Liver Function | Up to hour 168
  Liver function as measured by Total Bilirubin
Cardiovascular Function | Up to hour 168
  Cardiovascular function as measured by Mean arterial pressure. Scores less than 70 mmHg indicate worse outcomes.
State of Consciousness | Up to hour 168
  State of consciousness as measure by Glasgow Coma Scale which gives a score based on eye, verbal, and motor responses. Scores range from 3 to 15 with lower scores indicating worse outcome
Renal Function | Up to hour 168
  Renal function as measured by Creatinine.

CONTACTS AND LOCATIONS:
Locations (1):
- ShanghaiXinhua, Shanghai, China

IPD SHARING:
Plan to Share IPD: No